CLINICAL TRIAL: NCT07406503
Title: Modulation of the Stressed Brain: Effects of Transcranial Direct Current Stimulation on Stress Regulation and Episodic Future Thinking - an MRI Study in Healthy Volunteers
Brief Title: MRI-tDCS Stress and Future Thinking Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Sara De Witte, Dr., Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: tDCS FTS
Record Dates: First submitted 2025-11-26; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Healthy Participants
Keywords: tDCS; Episodic Future Thinking; Stress Regulation; MRI; fMRI; ASL; Spectroscopy; Cortisol; Mood

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Transcranial direct current stimulation (Active Comparator): Participants receive MRI-compatible transcranial direct current stimulation (tDCS) using a constant current of 2 mA applied for 20 minutes. The anodal electrode (4 × 4 cm) is positioned over the left dorsolateral prefrontal cortex (F3 position, neuronavigated) and the cathodal electrode over the contralateral orbitofrontal region. Stimulation is delivered while participants are in the MRI scanner.
  Interventions: Device: tDCS - Active non-invasive brain stimulation
- Sham Transcranial direct current stimulation (Placebo Comparator): Participants receive sham MRI-compatible transcranial direct current stimulation using the same electrode placement and setup as the active condition. The current is ramped up and down for approximately 30 seconds at the beginning of the session to mimic the initial sensation of stimulation, after which no current is delivered for the remainder of the 20-minute session. Stimulation is administered while participants are in the MRI scanner.
  Interventions: Device: tDCS - Sham non-invasive brain stimulation

INTERVENTIONS:
Device: tDCS - Active non-invasive brain stimulation — active non-invasive brain stimulation
  Arms: Active Transcranial direct current stimulation
Device: tDCS - Sham non-invasive brain stimulation — Sham non-invasive brain stimulation
  Arms: Sham Transcranial direct current stimulation

SUMMARY:
This academic study investigates how MRI-compatible transcranial direct current stimulation (tDCS) over the left dorsolateral prefrontal cortex (DLPFC) influences stress regulation and episodic future thinking in healthy volunteers. Participants undergo one MRI session: combining stress induction, tDCS (real or sham), and functional and metabolic MRI measurements. The study aims to better understand how non-invasive brain stimulation affects the neurophysiological and psychological mechanisms involved in stress processing and future-oriented thinking.

DETAILED DESCRIPTION:
The purpose of this study is to examine the modulatory effects of non-invasive brain stimulation on cognitive and emotional processes related to stress regulation and episodic future thinking (EFT).

Healthy adult volunteers complete one MRI session. Participants were randomly assigned to active or sham stimulation. First, participants performed an fMRI-based baseline measurement of the EFT task. This task involves imagining specific future personal events in response to cue words presented on a screen and later verbally describing these imagined events outside the scanner.

During the second part, participants complete the Montreal Imaging Stress Task (MIST) - a mental arithmetic paradigm with time pressure and negative feedback to induce acute stress. Immediately afterward, they receive MRI-compatible tDCS (active or sham) for 20 minutes while at rest. The active tDCS delivers 2 mA current through a 4×4 cm anode placed over the left DLPFC and a cathode over the contralateral orbitofrontal region. Sham stimulation follows the same setup with current ramping only at the onset and offset.

Following stimulation, an ASL perfusion scan, MRS spectroscopy targeting the hippocampus, and a post-stimulation EFT fMRI task were conducted. Throughout the MRI scan, behavioral and psychometric data were collected, including questionnaires on rumination, personality, and mood, as well as physiological and biochemical measures such as salivary cortisol and heart rate variability (HRV).

The primary goal is to assess whether active tDCS modulates the neural, endocrine, and behavioral correlates of stress and future-oriented cognition compared to sham stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-30 years.
* Right-handed, healthy volunteers.
* Native Dutch speakers with normal or corrected vision.
* No current or past psychiatric or neurological disorder.
* MRI-compatible (no metal implants, pacemaker, etc.).
* Not taking psychotropic medication.
* Provided written informed consent.

Exclusion Criteria:

* Pregnancy.
* History of epilepsy or neurosurgery.
* Cardiovascular, neurological, or severe medical illness.
* Claustrophobia or intolerance to MRI environment.
* Tattoos or piercings that cannot be removed.
* Alcohol or caffeine consumption within the restricted window before scanning.
* Current use of psychoactive substances or psychotropic drugs.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Specificity score of episodic future thinking | Baseline and immediately post-tDCS (single study visit)
  Specificity of episodic future thinking responses assessed using a standardized scoring procedure applied to imagined future events.
  Unit of Measure: EFT specificity score (units on a standardized scale)
Momentary mood ratings - fatigue | Baseline; immediately post-tDCS; and immediately post-EFT paradigm (single study visit)
  Self-reported tension measured using a visual analogue scale (VAS) Unit of Measure:Score on a 0-10 scale. A higher score means more fatigued.
Mean BOLD signal change during episodic future thinking | Baseline and immediately post-tDCS (single study visit)
  Mean blood-oxygen-level-dependent (BOLD) signal change during the episodic future thinking task, averaged across predefined prefrontal-limbic regions of interest.
  Unit of Measure: Percent signal change (or beta coefficients from the general linear model)
Momentary mood ratings -tension | Baseline; immediately post-tDCS; and immediately post-EFT paradigm (single study visit)
  Self-reported tension measured using a visual analogue scale (VAS) Unit of Measure: Score on a 0-10 scale. A higher score means more tensed.
Momentary mood ratings - vigor | Baseline; immediately post-tDCS; and immediately post-EFT paradigm (single study visit)
  Self-reported vigor measured using a visual analogue scale (VAS). Unit of Measure: Score on a 0-10 scale. A higher score means more vigor.
Momentary mood ratings - anger | Baseline; immediately post-tDCS; and immediately post-EFT paradigm (single study visit)
  Self-reported anger measured using a visual analogue scale (VAS). Unit of Measure: Score on a 0-10 scale. A higher score means more anger.
Momentary mood ratings - depressed mood | Baseline; immediately post-tDCS; and immediately post-EFT paradigm (single study visit)
  Self-reported depressed mood measured using a visual analogue scale (VAS). Unit of Measure: Score on a 0-10 scale. A higher score means more depressed mood.
Momentary mood ratings - cheerfulness | Baseline; immediately post-tDCS; and immediately post-EFT paradigm (single study visit)
  Self-reported cheerfulness measured using a visual analogue scale (VAS). Unit of Measure: Score on a 0-10 scale. A higher score means more cheerfulness.
Momentary mood ratings - stress | Baseline; immediately post-tDCS; and immediately post-EFT paradigm (single study visit)
  Self-reported stress measured using a visual analogue scale (VAS).
  Unit of Measure: Score on a 0-10 scale. A higher score means more stress.
Hippocampal glutamate concentration | Baseline and immediately post-tDCS (single study visit)
  Hippocampal glutamate concentration measured using proton magnetic resonance spectroscopy (¹H-MRS).
  Unit of Measure: Institutional units
Hippocampal GABA concentration | Baseline and immediately post-tDCS (single study visit)
  Hippocampal gamma-aminobutyric acid (GABA) concentration measured using proton magnetic resonance spectroscopy (¹H-MRS).
  Unit of Measure: Institutional units
Hippocampal glutamine concentration | Baseline and immediately post-tDCS (single study visit)
  Hippocampal glutamine concentration measured using proton magnetic resonance spectroscopy (¹H-MRS).
Hippocampal N-acetylaspartate (NAA) concentration | Baseline and immediately post-tDCS (single study visit)
  Hippocampal N-acetylaspartate (NAA) concentration measured using proton magnetic resonance spectroscopy (¹H-MRS).
  Unit of Measure: Institutional units

SECONDARY OUTCOMES:
Salivary cortisol concentration | Baseline, immediately post-tDCS, and immediately post-EFT task (single study visit)
  Salivary cortisol concentration measured using biochemical assay from saliva samples.
  Unit of Measure: nmol/L (or µg/dL)
Cerebral blood flow | Baseline and Periprocedural (during tDCS)
  Cerebral blood flow measured using arterial spin labeling (ASL) MRI. Unit of Measure: mL/100 g/min

OTHER OUTCOMES:
Depressive symptom severity | Baseline (prior to any intervention)
  Beck Depression Inventory (BDI-II) The BDI-II consists of 21 items, each scored 0-3. Unit of Measure: BDI-II total score ranging from 0 to 63. Higher scores indicate more depressive symptoms.
Body mass index | Baseline (prior to any intervention)
  Body mass index calculated from measured body weight and height.
Trait rumination | Baseline (prior to any intervention)
  Trait rumination assessed using the Ruminative Responses Scale (RRS). Unit of Measure: RRS total score (range 22-88; higher scores indicate greater trait rumination).
Brooding rumination | Baseline (single study visit)
  Brooding rumination assessed using the Brooding subscale of the Ruminative Responses Scale (BSRI).
  Unit of Measure: BSRI (Brooding) subscale score, range 5-20; higher scores indicate greater brooding rumination.
Trait anxiety | Baseline (single study visit)
  Trait anxiety assessed using the State-Trait Anxiety Inventory, Trait version (STAI-T).
  Unit of Measure: STAI-T total score (range 20-80; higher scores indicate greater trait anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No